CLINICAL TRIAL: NCT02658006
Title: Evaluation of Multimodal Monitoring Technologies in the Peri-operative Care of Cardiac Surgical Patients
Brief Title: Evaluation of Monitoring TECHNOlogies in the PERI-OPerative Care of Cardiac Surgical Patients
Acronym: TechnoPeriOp
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Andre Denault, MD PhD FRCPC ABIM-CCM, Montreal Heart Institute
Other Study IDs: 2015-1903
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: C.Surgical Procedure; Cardiac; Right-Sided Heart Failure; Acute Kidney Injury; Respiratory Insufficiency; Postoperative Complications
Keywords: Near Infrared Spectroscopy; Ultrasonography; Hepatic vein Doppler; Portal vein Doppler; Lung ultrasound; Positive fluid balance; Mixed venous saturation
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury; Respiratory Insufficiency; Postoperative Complications | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgical patients: Adult patients having a cardiac surgery at the Montreal Heart Institute
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — All cardiac surgery procedures

SUMMARY:
The purpose of this prospective observational cohort study is to evaluate multimodal monitoring technologies in the perioperative care of cardiac surgical patients. Right ventricular pressure tracings, near infrared spectroscopy (NIRS) and transthoracic ultrasonography will be studied for their ability to detect and predict complications such as right ventricular failure, renal failure and respiratory failure.

DETAILED DESCRIPTION:
The study has 4 main objectives:

1. To determine if right ventricular pressure tracings correlate with other indices of right ventricular failure and with positive fluid balance, renal failure and increased length of stay in the intensive care unit.
2. To determine the prevalence of portal vein pulsatility in the perioperative period and its association with right ventricular failure and positive fluid balance.
3. To determine if Near InfraRed Spectroscopy (NIRS) values correlate with mixed venous oxygen saturation (SvO2) and with poorer post-operative prognosis.
4. To determine the incidence, risk factors and prognosis of respiratory complications of cardiac surgery using transthoracic ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery performed at the Montreal Heart Institute
* 18 years old and older

Exclusion Criteria:

* Urgent surgery
* Pre-operative intra-aortic balloon pump, left ventricular assist device or ECMO
* Heart transplant
* Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having any cardiac surgery at the Montreal Heart Institute.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Right ventricular failure | First 24 hours post cardiac surgery
Pulmonary complications | 30 days
  Composite outcome : pneumonia, prolonged mechanical ventilation (more than 24 hours) or clinically significant atelectasis (requiring > 2L O2).
Acute Renal failure | 30 days
  KDIGO : class I and more

SECONDARY OUTCOMES:
Fluid balance | First 24h
Maximal blood lactate levels | First 24h

CONTACTS AND LOCATIONS:
Overall Officials: André Y Denault, MD, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denault A, Lamarche Y, Rochon A, Cogan J, Liszkowski M, Lebon JS, Ayoub C, Taillefer J, Blain R, Viens C, Couture P, Deschamps A. Innovative approaches in the perioperative care of the cardiac surgical patient in the operating room and intensive care unit. Can J Cardiol. 2014 Dec;30(12 Suppl):S459-77. doi: 10.1016/j.cjca.2014.09.029. Epub 2014 Oct 5. PMID 25432139
- [Background] Prowle JR, Echeverri JE, Ligabo EV, Ronco C, Bellomo R. Fluid balance and acute kidney injury. Nat Rev Nephrol. 2010 Feb;6(2):107-15. doi: 10.1038/nrneph.2009.213. Epub 2009 Dec 22. PMID 20027192
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: II. Pathophysiology, clinical importance, and management. Anesth Analg. 2009 Feb;108(2):422-33. doi: 10.1213/ane.0b013e31818d8b92. PMID 19151265
- [Background] McNaughton DA, Abu-Yousef MM. Doppler US of the liver made simple. Radiographics. 2011 Jan-Feb;31(1):161-88. doi: 10.1148/rg.311105093. PMID 21257940
- [Background] Catalano D, Caruso G, DiFazzio S, Carpinteri G, Scalisi N, Trovato GM. Portal vein pulsatility ratio and heart failure. J Clin Ultrasound. 1998 Jan;26(1):27-31. doi: 10.1002/(sici)1097-0096(199801)26:13.0.co;2-l. PMID 9475205
- [Background] Zheng F, Sheinberg R, Yee MS, Ono M, Zheng Y, Hogue CW. Cerebral near-infrared spectroscopy monitoring and neurologic outcomes in adult cardiac surgery patients: a systematic review. Anesth Analg. 2013 Mar;116(3):663-76. doi: 10.1213/ANE.0b013e318277a255. Epub 2012 Dec 24. PMID 23267000
- [Background] Nagdyman N, Ewert P, Peters B, Miera O, Fleck T, Berger F. Comparison of different near-infrared spectroscopic cerebral oxygenation indices with central venous and jugular venous oxygenation saturation in children. Paediatr Anaesth. 2008 Feb;18(2):160-6. doi: 10.1111/j.1460-9592.2007.02365.x. PMID 18184248
- [Background] Afilalo J, Eisenberg MJ, Morin JF, Bergman H, Monette J, Noiseux N, Perrault LP, Alexander KP, Langlois Y, Dendukuri N, Chamoun P, Kasparian G, Robichaud S, Gharacholou SM, Boivin JF. Gait speed as an incremental predictor of mortality and major morbidity in elderly patients undergoing cardiac surgery. J Am Coll Cardiol. 2010 Nov 9;56(20):1668-76. doi: 10.1016/j.jacc.2010.06.039. PMID 21050978
- [Background] Weissman C. Pulmonary complications after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2004 Sep;8(3):185-211. doi: 10.1177/108925320400800303. PMID 15375480
- [Background] Lobo V, Weingrow D, Perera P, Williams SR, Gharahbaghian L. Thoracic ultrasonography. Crit Care Clin. 2014 Jan;30(1):93-117, v-vi. doi: 10.1016/j.ccc.2013.08.002. PMID 24295842
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Derived] Cavayas YA, Eljaiek R, Rodrigue E, Lamarche Y, Girard M, Wang HT, Levesque S, Denault AY. Preoperative Diaphragm Function Is Associated With Postoperative Pulmonary Complications After Cardiac Surgery. Crit Care Med. 2019 Dec;47(12):e966-e974. doi: 10.1097/CCM.0000000000004027. PMID 31609771
- [Derived] Eljaiek R, Cavayas YA, Rodrigue E, Desjardins G, Lamarche Y, Toupin F, Denault AY, Beaubien-Souligny W. High postoperative portal venous flow pulsatility indicates right ventricular dysfunction and predicts complications in cardiac surgery patients. Br J Anaesth. 2019 Feb;122(2):206-214. doi: 10.1016/j.bja.2018.09.028. Epub 2018 Nov 28. PMID 30686306